CLINICAL TRIAL: NCT03219034
Title: Mid-line Traction Versus Bilateral Thrust Oral Appliances: A Trial to Determine Superiority for Improving Upper Airway Function and Sleep Quality
Brief Title: Trial on Oral Appliance Design for Improving Upper Airway Function and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Emet D. Schneiderman, PhD, Professor Dr., Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0390
Record Dates: First submitted 2017-07-11; First posted 2017-07-17 (Actual); Results first posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: oral appliance; sleep quality; sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Oral appliance - A (Experimental): Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth and uses a Midline Traction Mechanism to advance the mandible. The coupling mechanism is located at a single point midline, allows adjustment by incremental protraction (advancement) of the mandible.
  Trade Name: "TAP1" Oral Appliance, Airway Management Inc. Dallas, TX
  Interventions: Device: oral appliance - A ; washout; oral appliance B; Device: oral appliance - B; washout; oral appliance A
- Oral appliance - B (Experimental): Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth uses a Bilateral Thrust Mechanism to advance the mandible. The trays are engaged by means of adjustable lugs.
  Trade name: "SomnoDent Flex" Oral Appliance, SomnoMed Inc., Plano TX
  Interventions: Device: oral appliance - A ; washout; oral appliance B; Device: oral appliance - B; washout; oral appliance A

INTERVENTIONS:
Device: oral appliance - A ; washout; oral appliance B — Anti-snoring intra-oral appliance A that consists of two custom fitted trays which fit over the upper and lower teeth and uses a Midline Traction Mechanism to advance the mandible. The coupling mechanism is located at a single point midline, allows adjustment by incremental protraction (advancement) of the mandible. 1 week washout followed by anti-snoring intra-oral appliance B that consists of two custom fitted trays which fit over the upper and lower teeth uses a Bilateral Thrust Mechanism to advance the mandible. The trays are engaged by means of adjustable lugs.
  Other Names: "TAP1" Oral Appliance; washout; "SomnoDent Flex"
Device: oral appliance - B; washout; oral appliance A — Anti-snoring intra-oral appliance B that consists of two custom fitted trays which fit over the upper and lower teeth uses a Bilateral Thrust Mechanism to advance the mandible. The trays are engaged by means of adjustable lugs. 1-week washout followed by anti-snoring intra-oral appliance A that consists of two custom fitted trays which fit over the upper and lower teeth and uses a Midline Traction Mechanism to advance the mandible. The coupling mechanism is located at a single point midline, allows adjustment by incremental protraction (advancement) of the mandible.
  Other Names: "SomnoDent Flex"; washout; "TAP1"

SUMMARY:
This study will compare the effectiveness of the two leading oral appliances (OAs) designs for the treatment of severe obstructive sleep apnea in overweight adults. The effectiveness of OAs has come under question since different designs are combined in evaluating treatment efficacy, for example when comparing them to continuous positive airway pressure Due to the wide range of reported efficacy (53 to 90%), it is of great value to identify the most effective design to guide sleep practitioners and patients.

DETAILED DESCRIPTION:
The two prominent oral appliances used in treating obstructive sleep apnea differ in their designs, mid-line traction versus bilateral thrust. From a clinical perspective, it is important to know which design is superior and should be the 'treatment of choice' for improving airway function and sleep quality. These two designs differ in their protrusive mechanisms that are categorized in general under four main types: bilateral compression, bilateral thrust, midline compression and mid-line traction. Although the two designs considered in this proposal have undergone the most rigorous testing individually, well controlled 'head-to-head' trials as proposed here have not been conducted to determine their efficacy within a single test population.

ELIGIBILITY:
Inclusion Criteria:

* OSA PSG or PG diagnosed adults within 1 year
* age >18
* Currently treated with continuous positive airway pressure (CPAP)
* AHI ≥ >30 events/hour of sleep
* Two or more OSA symptoms (snoring, witnessed apnea or daytime hypersomnolence complaint)
* BMI ≥ 30
* At least 8 teeth per arch to support either OA device
* Central and mixed apnea index <5 events/hour
* Mallampati score from I to III
* Palatine tonsils - grade 0, 1, or 2
* Consent to study's timeline
* Willingness to wear home sleep test apparatus for at least 4 nights
* Willingness to wear an oral appliance every night for 8 weeks
* Willingness to pick up and return home sleep test kits as needed

Exclusion Criteria:

* Cardiac & pulmonary disease (e.g., congestive heart failure, severe arrhythmias, COPD);
* Central sleep apnea;
* Comorbidities with other sleep disorders
* No active TMD or jaw muscle pain
* Morphological airway abnormalities
* Pre-existing difficulty swallowing; throat or neck related health issues
* Endocrine dysfunction
* Severe psychiatric disorders;
* Previous OA therapy; ENT surgery
* Restrictions in jaw opening
* Pregnancy / breast feeding or intent to become pregnant during the study
* Inability to apply the sleep recorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emet Schneiderman, PhD, Principal Investigator — Texas A&M University College of Dentistry
Locations (1):
- Texas A&M University College of Dentistry, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schneiderman E, Schramm P, Hui J, Wilson PD, Moura P, German Z, McCann A, Newton M. Randomized Trial of 2 Self-Titrated Oral Appliances for Airway Management. J Dent Res. 2021 Feb;100(2):155-162. doi: 10.1177/0022034520956977. Epub 2020 Sep 18. PMID 32942939

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 162 individuals screened for eligibility; 62 enrolled.
Groups:
- Oral Appliance Sequence A-B: Group STARTING with Appliance A for 4 weeks: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth and uses a Midline Traction Mechanism to advance the mandible. The coupling mechanism is located at a single point midline, allows adjustment by incremental protraction (advancement) of the mandible. Used for period of first 4 weeks.
  Trade Name: "TAP1" Oral Appliance, Airway Management Inc. Dallas, TX
  Used Appliance B for second leg of 4 weeks: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth uses a Bilateral Thrust Mechanism to advance the mandible. The trays are engaged by means of adjustable lugs.
  Trade name: "SomnoDent Flex" Oral Appliance, SomnoMed Inc., Plano TX
- Oral Appliance Sequence B-A: Group STARTING with Appliance B for 4 weeks: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth uses a Bilateral Thrust Mechanism to advance the mandible. The trays are engaged by means of adjustable lugs.
  Trade name: "SomnoDent Flex" Oral Appliance, SomnoMed Inc., Plano TX
  Used Appliance A for second leg of 4 weeks: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth and uses a Midline Traction Mechanism to advance the mandible. The coupling mechanism is located at a single point midline, allows adjustment by incremental protraction (advancement) of the mandible. Used for period of first 4 weeks.
  Trade Name: "TAP1" Oral Appliance, Airway Management Inc. Dallas, TX
Period: Overall Study
Arm/Group | Oral Appliance Sequence A-B | Oral Appliance Sequence B-A
Started | 31 | 31
Completed | 20 | 16
Not Completed | 11 | 15
Not completed — Lost to Follow-up | 9 | 13
Not completed — Additional dental work needed | 1 | 0
Not completed — UPPP Surgery | 1 | 0
Not completed — Dental sensitivity | 0 | 1
Not completed — Death in family | 0 | 1

BASELINE CHARACTERISTICS:
Population: 31 subjects assigned to each oral appliance (OA) sequence group in cross-over design. 6 left study prior to receipt of OA, so demographics reflect those 56 subjects who received the intervention. See figure 1 in publication for details.
Groups:
- Oral Appliance Sequence - A -- B: Group STARTING with Appliance A for 4 weeks: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth and uses a Midline Traction Mechanism to advance the mandible. The coupling mechanism is located at a single point midline, allows adjustment by incremental protraction (advancement) of the mandible. Trade Name: "TAP1" Oral Appliance, Airway Management Inc. Dallas, TX. One week washout with no oral appliance usage.
  Used Appliance B for second leg of 4 weeks: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth uses a Bilateral Thrust Mechanism to advance the mandible. The trays are engaged by means of adjustable lugs. Trade name: "SomnoDent Flex" Oral Appliance, SomnoMed Inc., Plano TX.
- Oral Appliance Sequence B -- A: Group STARTING with Appliance B for first leg of 4 weeks: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth uses a Bilateral Thrust Mechanism to advance the mandible. The trays are engaged by means of adjustable lugs. Trade name: "SomnoDent Flex" Oral Appliance, SomnoMed Inc., Plano TX. One week washout with no oral appliance usage.
  Used Appliance A for second leg of 4 weeks: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth and uses a Midline Traction Mechanism to advance the mandible. The coupling mechanism is located at a single point midline, allows adjustment by incremental protraction (advancement) of the mandible. Trade Name: "TAP1" Oral Appliance, Airway Management Inc. Dallas, TX
- Total: Total of all reporting groups
Arm/Group | Oral Appliance Sequence - A -- B | Oral Appliance Sequence B -- A | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.5 [46.3 to 69.0] | 61.0 [52.0 to 66.0] | 61.0 [51.0 to 68.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 15 | 24 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 21 | 22 | 43
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (kg/m^2) [Median (Inter-Quartile Range); unit: kg/m^2] | 30.3 [27.4 to 34.0] | 31.0 [28.0 to 33.6] | 31.0 [29.9 to 33.8]
Respiratory Event Index (events/hr) [Median (Inter-Quartile Range); unit: number of events /hour] — Number of respiratory events per hour (number of apnea-hypopnea events divided by the number of recorded hours)
  number of events /hour | 32.6 [17.9 to 41.8] | 36.1 [22.3 to 57.9] | 33.7 [20.7 to 54.9]
Mean SaO2 [Median (Inter-Quartile Range); unit: Percent] — Mean percentage of oxygen saturation values were obtained from each subject using pulse oximetry. Collectively these were not normally distributed so were summarized with the median and interquartile range.
  Percent | 93.0 [92.0 to 94.6] | 93.1 [91.0 to 95.4] | 93.0 [91.0 to 95.0]
Minimum SaO2 [Median (Inter-Quartile Range); unit: Percent] — Minimum oxygen percentage saturation values were obtained for each subject using pulse oximetry. Collectively these were not normally distributed so were summarized with the median and interquartile range.
  Percent | 80.0 [76.0 to 85.0] | 82.0 [77.0 to 87.0] | 80.0 [77.0 to 85.0]

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Event Index (REI) at T2
Description: Number of apneas and hypopneas (respiratory events) per hour of recording; REI was reported instead of AHI, as it is a more appropriate measure for home sleep testing.
Time Frame: 4 weeks
Population: 20 subjects dropped out or were lost to follow-up by T2. An additional 6 dropped out before T4, bringing the total number of dropouts to 26.
Measure: Median (Inter-Quartile Range); unit: number of events per hour
Groups:
- Oral Appliance Sequence - A -- B: Group STARTING with this appliance: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth and uses a Midline Traction Mechanism to advance the mandible. The coupling mechanism is located at a single point midline, allows adjustment by incremental protraction (advancement) of the mandible.
  Trade Name: "TAP1" Oral Appliance, Airway Management Inc. Dallas, TX.
  1 week washout followed by Appliance B for 4 weeks: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth uses a Bilateral Thrust Mechanism to advance the mandible. The trays are engaged by means of adjustable lugs.
  Trade name: "SomnoDent Flex" Oral Appliance, SomnoMed Inc., Plano TX
- Oral Appliance Sequence B -- A: Group STARTING with Appliance B for 4 weeks: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth uses a Bilateral Thrust Mechanism to advance the mandible. The trays are engaged by means of adjustable lugs.
  Trade name: "SomnoDent Flex" Oral Appliance, SomnoMed Inc., Plano TX Used Appliance A for second leg of 4 weeks: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth and uses a Midline Traction Mechanism to advance the mandible. The coupling mechanism is located at a single point midline, allows adjustment by incremental protraction (advancement) of the mandible. Used for period of first 4 weeks.
  Trade Name: "TAP1" Oral Appliance, Airway Management Inc. Dallas, TX
Arm/Group | Oral Appliance Sequence - A -- B | Oral Appliance Sequence B -- A
Number analyzed (Participants) | 21 | 21
number of events per hour
  At T2 (end of 1st 4 wk leg | 12.8 [7.5 to 26.7] | 21.1 [9.8 to 31.2]
  At T4 (end of 2nd 4 wk leg): number analyzed (Participants) | 20 | 16
  At T4 (end of 2nd 4 wk leg) | 9.3 [7.7 to 15.5] | 13.1 [10.4 to 16.6]
Statistical Analysis 1: Comparison: Oral Appliance Sequence - A -- B vs Oral Appliance Sequence B -- A; Cross-over design: Median differences between oral appliances at the end of the first 4-week leg of the study (T2). The hypothesis tested was that REI would be lowered more with Appliance A than B; Test type: Superiority; p = 0.152, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 3.8

2. Secondary Outcome: Stable Sleep Percent
Description: Percent of stable sleep during the recording, specifically the percentage of high frequency coupling (HFC%) from cardiopulmonary coupling (CPC) Analysis
Time Frame: 4 weeks
Population: 20 subject dropped out or were lost to follow-up at T2. An additional 6 dropped out before T4.
Measure: Mean (Standard Deviation); unit: percentage of high frequency coupling
Groups:
- Oral Appliance Sequence - A -- B: Group STARTING with this appliance: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth and uses a Midline Traction Mechanism to advance the mandible. The coupling mechanism is located at a single point midline, allows adjustment by incremental protraction (advancement) of the mandible.
  Trade Name: "TAP1" Oral Appliance, Airway Management Inc. Dallas, TX
- Oral Appliance Sequence B-A: Group STARTING with this appliance: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth uses a Bilateral Thrust Mechanism to advance the mandible. The trays are engaged by means of adjustable lugs.
  Trade name: "SomnoDent Flex" Oral Appliance, SomnoMed Inc., Plano TX
Arm/Group | Oral Appliance Sequence - A -- B | Oral Appliance Sequence B-A
Number analyzed (Participants) | 21 | 21
percentage of high frequency coupling
  At T2 (end of 1st 4 wk leg | 49.35 (17.70) | 48.7 (18.3)
  At T4 (end of 2nd 4 wk leg: number analyzed (Participants) | 20 | 16
  At T4 (end of 2nd 4 wk leg | 47.82 (21.12) | 52.38 (19.67)

ADVERSE EVENTS:
Time Frame: Each participant participated for 9 weeks, for which time adverse event data were collected.
Groups:
- Oral Appliance A: Oral Appliance A - Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth and uses a Midline Traction Mechanism to advance the mandible. The coupling mechanism is located at a single point midline, allows adjustment by incremental protraction (advancement) of the mandible. Trade Name: "TAP1" Oral Appliance, Airway Management Inc. Dallas, TX. Worn for 4 weeks.
- Oral Appliance B: Oral Appliance B: Anti-snoring intra-oral appliance that consists of two custom fitted trays which fit over the upper and lower teeth uses a Bilateral Thrust Mechanism to advance the mandible. The trays are engaged by means of adjustable lugs. Trade name: "SomnoDent Flex" Oral Appliance, SomnoMed Inc., Plano TX. Worn for 4 weeks.
Arm/Group | Oral Appliance A | Oral Appliance B
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/36
Other Adverse Events (participants affected / at risk) | 0/41 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Appliance A (N=41) | Oral Appliance B (N=36)
Oral appliance intolerance (General disorders) | 0 | 1 — Intolerance to oral appliance therapy due to dental sensitivity. This occurred in a subject in Sequence B-A in response to oral appliance B during the first leg of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03219034/Prot_SAP_001.pdf
  • Informed Consent Form (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03219034/ICF_002.pdf